CLINICAL TRIAL: NCT05518435
Title: Managing Young People With Attention Deficit Hyperactivity Disorder in Primary Care (MAP) Study: Mapping Current Practice and Co-producing Guidance to Improve Healthcare in an Underserved Population
Brief Title: Managing Young People With ADHD in Primary Care Study
Acronym: MAP
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 313424; MHF008 (Other Grant/Funding Number: National Institute for Health and Care Research)
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: ADHD
Keywords: Young adult; Service provision
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Observation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Work package 1 (WP1) - survey: WP1 aims to recruit a minimum of 252 survey respondents, providing a minimum of six responses for each of the 42 Integrated Care Systems (ICSs) in England. The aim will be to gather responses from as many respondents as possible, to provide as much information as possible on primary care provision across over >1200 PCNs in England. This will provide the first national overview of prescribing practice and the availability of health care for young people with ADHD through primary care in England. The inclusion of three stakeholder groups (health professional, service users, and commissioners/providers) will ensure that the survey includes reports from a balance of perspectives and provide the opportunity to compare data between groups and locations.
  The sampling frame for WP1 includes all stakeholders aged 16 or over with an interest in providing or receiving health care for young people with ADHD, as well as those involved in providing/commissioning local primary care provision.
  Interventions: Other: None, observational study
- Work package 2 (WP2) - qualitative study: WP2 aims to recruit between 20 and 30 participants, consisting of 10-15 young people (aged 16-25) with ADHD and their parent carers and 10-15 health professionals and commissioners/providers. Participants will be recruited from between three and six geographic locations (e.g., PCNs), dependent on findings from WP1. This sample size will enable qualitative data to be collected from approximately five participants per location.
  The sampling frame for WP2 consists of a purposive selection of stakeholders.
  Interventions: Other: None, observational study
- Work package 3 (WP3) - co-production of guidance: WP3 aims to recruit between six and 16 participants, consisting of 2-6 young people (aged 16-25) with ADHD and/or their parents/carers, 2-6 health professional and/or commissioners/providers, and between 1 and 4 members of the research team. The sample will be sufficient to include perspectives from identified key stakeholders, while the relatively small group size will support close group work. The small sample size will also enable delivery of key features of co-production research such as building strong relationships and providing opportunities for growth and development of participants.
  The sampling frame for WP3 consists of a purposive selection of key stakeholders. In addition to the key stakeholder groups outlined above, co-production activities will also involve MAP study researchers.
  Interventions: Other: None, observational study

INTERVENTIONS:
Other: None, observational study — The MAP study involves mapping current practice (WP1), exploring current experiences (WP2), and co-creating guidance based on existing evidence (WP3).

SUMMARY:
Background:

Attention deficit hyperactivity disorder (ADHD) is the most common childhood neurodevelopmental disorder. It affects around 5% of children and adolescents, and up to 40% continue to experience symptoms into adulthood. Primary care practitioners (e.g., general practitioners (GPs), nurses, link workers, clinical pharmacists) play an important role in the healthcare of young people (YP) with ADHD, particularly due to long waiting times in adult mental health services, and patchy provision of specialist services. However, many practitioners feel unsure about how to support YP at this vulnerable stage in their lives. Practitioners report concerns about prescribing ADHD medication and a desire for more guidance. Currently, little is known about how YP with ADHD are supported in primary care, the strengths and weakness of existing care pathways, and how care can be improved.

Aims:

To provide an evidence-base by mapping current services, and co-produce guidance to improve and better co-ordinate primary care for YP aged 16-25 with ADHD.

Methods:

Three interlinked studies. A mapping study including a national survey of stakeholders to map patient pathways, prescribing practice, shared-care arrangements, and practitioner roles. A qualitative study including semi-structured interviews with YP and practitioners, to gain insight into experiences of 'what works' and 'what is needed'. Workshops to co-develop a map of patient pathways, key messages, and clinical guidance.

Patient Involvement:

This research has been developed in response to identified gaps in services, and requests from people with ADHD. The team includes young people with ADHD whose input will help ensure the research is sensitive and relevant, and an academic GP to ensure identified solutions are deliverable within primary care settings.

Impact:

The expected impact of this research is improvement of the quality and experience of care for YP with ADHD. Also, to improve experiences of primary care providers facing difficulties managing ADHD.

DETAILED DESCRIPTION:
This research aims to map current services and co-create evidence-based guidance to improve and better co-ordinate primary care for young people aged 16-25 years with ADHD.

OBJECTIVES

The objectives of this research are to:

1. Develop a national map and overview of current primary care pathways and prescribing practice in the management of young people with ADHD
2. Explore:

   1. Primary care providers and related organisations' needs for information resources and prescribing support in their roles managing care for young people with ADHD
   2. The expectations and needs of young people aged 16-25 regarding primary care ADHD support, information, and management
3. Co-produce evidence informed guidance to better co-ordinate primary care for young people with ADHD, based on discussions around findings from objectives 1, 2a and 2b

OUTCOMES

The outcomes of this research will be shaped by close work with professionals and members of the community, via the practice and policy research advisory group (P-RAG) and young person and parent/carer research advisory group (Y-RAG) groups, to ensure their relevance and utility. Anticipated outcomes include:

1. National overview of primary care provision for young people with ADHD across England, including:

   1. Geographic map, showing variation in provision by NHS region or appropriate organisational boundaries
   2. Summary of existing care pathways for the management of young people with ADHD in primary care, including exemplars of best practice
2. Qualitative summary of the perspectives of people involved in delivering and in need of care, on the management of ADHD in primary care including:

   1. Health professionals' needs for information resources and prescribing support
   2. Young people with ADHD and their parent/carers' needs for information resources, healthcare, and support with self-management
3. Co-produced guidance on how to better co-ordinate and design primary care for young people aged 16-25 with ADHD.

STUDY DESIGN and METHODS Overview: This mixed methods study consists of three work packages. Each WP involves data collection/creation working with the following stakeholder groups.

* Patients, with a focus on young people (aged 16-25) with ADHD, and their parent/carers
* Health professionals, with a focus on those in primary care (including general practitioners (GPs), specialist nurses, mental health practitioners, and clinical pharmacists)
* Commissioners/providers of NHS healthcare for people with ADHD

ELIGIBILITY:
Participants will include people aged 16 or over with lived experience of ADHD (and their parent/carers), health professionals with a focus on primary care (such as GPs, nurses, mental health practitioners, and clinical pharmacists), and primary care commissioners/providers. Sampling, recruitment strategies, and eligibility criteria, vary slightly between work packages, as outlined below.

WP1 SURVEY

Inclusion Criteria:

Self-identifies as

* Being at least one of the following:

  * A person aged 16 or over with lived experience of ADHD, or parent/carer of a person with ADHD
  * Health professional (person working in any role that provides healthcare services, include NHS, voluntary and private services, clinical, managerial, leadership and administrative roles)
  * Commissioner/provider of National Health Service (NHS) healthcare services (e.g., member of clinical commissioning group, primary care network (PCN), integrated care system (ICS), or another NHS organisation)
* Currently resident, working, or studying in England

Exclusion Criteria:

* Does not identify as a person aged 16 or over with lived experience of ADHD, a health professional, or a commissioner/provider of NHS health services
* Not currently resident, working, or studying in England

WP2 QUALITATIVE STUDY

Inclusion Criteria:

* One of the following:

  * Young person aged 16-25 with lived experience of ADHD, or a parent/carer of a young person with ADHD
  * Health professional (person that provides healthcare services with a focus on primary care, including clinical, managerial, leadership and administrative roles)
  * Commissioner/provider of healthcare services (e.g., member of clinical commissioning group, PCN, ICS, NHS, or another organisation)
* Currently resident or working in England
* Currently resident or working close to one of the qualitative study sites identified following WP1, where 'close to' means located within the same geographic locality (to be decided based on findings from WP1)

Exclusion Criteria:

* Not a young person aged 16-25 with lived experience of ADHD (or a parent/carer), a health professional, or commissioner/provider of health services
* Not currently resident or working in England
* Not currently resident, working, or studying close to one of the qualitative study sites identified following WP1, where 'close to' means located within the same geographic locality (to be decided based on findings from WP1)

WP3 Co-PRODUCTION

Inclusion Criteria:

* One of the following:

  * Young person aged 16-25 with lived experience of ADHD, or a parent/carer of a young person with ADHD
  * Health professional (person that provides healthcare services, including clinical, managerial, leadership and administrative roles)
  * Commissioner/provider of NHS healthcare services (e.g., member of clinical commissioning group, PCN, ICS, local authority, or another NHS organisation)
  * A member of the MAP study research team
* Currently resident, working, or studying in England
* Willing and able to work collaboratively and engage in consultations to co-produce evidence-based guidance for improving the co-ordination of primary care for young people with ADHD

Exclusion Criteria:

* Not a young person aged 16-25 with lived experience of ADHD (or a parent/carer), a health professional, commissioner/provider of NHS health services, or a member of the MAP study research team
* Not currently resident, working, or studying in England
* Not willing and able to work collaboratively and engage in consultations to co-produce evidence-based guidance for improving the co-ordination of primary care for young people with ADHD

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: WP1 SURVEY The sampling frame for WP1 includes all stakeholders aged 16 or over with an interest in providing or receiving health care for young people with ADHD, as well as those involved in providing/commissioning local primary care provision.
  WP2 QUALITATIVE STUDY The sampling frame for WP2 consists of a purposive selection of stakeholders.
  WP3 CO-PRODUCTION The sampling frame for WP3 consists of a purposive selection of key stakeholders. In addition to the key stakeholder groups outlined above, co-production activities will also involve MAP study researchers.
Sampling Method: Non-Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
WP1: Reports of the prescribing of adult ADHD medication, by primary care practices in England | At time of completing survey
  WP1 (national survey) will report on prescribing of ADHD medication by primary care practices in England. Outcome data will be communicated as a summary total of 'yes' / 'no' survey responses, and analysed by the geographic location of practices, as well as the type of respondent reporting this practice (e.g., person with ADHD, clinician, or commissioner)

SECONDARY OUTCOMES:
WP1: Reports of shared care agreements being in place for prescribing of adult ADHD medication, by local primary care practices (in England) | At time of completing survey
  WP1 (national survey) will report on the presence of shared care agreements for prescribing of ADHD medication by primary care practices in England. Outcome data will be communicated as a summary total of 'yes' / 'no' survey responses, and analysed by the geographic location of practices, as well as the type of respondent reporting this practice (e.g., person with ADHD, clinician, or commissioner)
WP1: Reports of mental health support being in place for patients with adult ADHD medication, by local primary care practices (in England) | At time of completing survey
  WP1 (national survey) will report on the presence of shared care agreements for prescribing of ADHD medication by primary care practices in England. Outcome data will be communicated as a summary total of 'yes' / 'no' survey responses, and analysed by the geographic location of practices, as well as the type of respondent reporting this practice (e.g., person with ADHD, clinician, or commissioner)
WP2: Qualitative summary of the perspectives of people involved in delivering and in need of care, on the management of ADHD in primary care medication, by local primary care practices (in England) | At time of interview
  WP2 (qualitative study) will report on experiences of primary care provision for young people with ADHD across England, from the perspectives of health professionals and young people with ADHD. Topics covered will include, prescribing practice, shared care agreements, and information provision.

OTHER OUTCOMES:
WP3: Co-produced guidance on how to better co-ordinate and design primary care for young people aged 16-25 with ADHD. | At time of co-production workshops
  WP3 (co-production study) will deliver an output in the form of co-produced guidance on how to better co-ordinate and design primary care for young people aged 16-25 with ADHD.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Price, PhD, Principal Investigator — University of Exeter Medical School
Locations (1):
- Anna Price, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Arrangements for access to the final study dataset are outlined in the MAP study data management plan. In summary:
  * Only members of the study research team will have access to the full dataset.
  * It is possible that anonymised data from this dataset may be used for secondary analysis. This possibility is detailed in the study Participant Information Sheet (PIS) and Consent forms and would therefore only take place with the consent of the participants. All patient documentation reflects the possible future use an anonymised subset of these data in research.

REFERENCES:
- [Derived] Price A, Smith JR, Mughal F, Salimi A, Melendez-Torres GJ, Newlove-Delgado T. Protocol for the mixed methods, Managing young people (aged 16-25) with Attention deficit hyperactivity disorder in Primary care (MAP) study: mapping current practice and co-producing guidance to improve healthcare in an underserved population. BMJ Open. 2023 Jul 10;13(7):e068184. doi: 10.1136/bmjopen-2022-068184. PMID 37429692
- See also: Study website, with additional background information. Public facing, and hosted by Sponsor organisation (University of Exeter) — https://sites.exeter.ac.uk/mapadhd/